CLINICAL TRIAL: NCT07402915
Title: An Open-label, Fixed Sequence Phase I Study to Evaluate the Effect of Itraconazole (a Strong CYP3A Inhibitor) on the Pharmacokinetics of AZ14170132, the TOP1 Inhibitor Payload of the Antibody Drug Conjugate AZD5335, in Participants With Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Brief Title: Drug-drug Interaction Study With AZD5335 and Itraconazole in Participants With Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D8991C00002; EU CT (Other: 2025-522731-34-00)
Record Dates: First submitted 2026-01-23; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal
Keywords: CYP3A inhibitor; TOP1 inhibitor payload
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD5335/AZD5335 + Itraconazole (Experimental): In Part A, participants will receive AZD5335 alone as an intravenous (IV) infusion, and in combination with oral itraconazole, every 3 weeks (Q3W) from cycle 1 to cycle 3. In Part B, participants will receive AZD5335 as an IV infusion Q3W, from Day 1 of Cycle 4 until progression, unacceptable toxicity or any other specified criteria for discontinuation occurs.
  Interventions: Drug: AZD5335; Drug: Itraconazole

INTERVENTIONS:
Drug: AZD5335 — AZD5335 will be administered as IV infusion.
  Other Names: AZ14170132
Drug: Itraconazole — Itraconazole capsule will be administered orally.

SUMMARY:
The purpose of this study is to assess the effect of itraconazole on the pharmacokinetics (PK) of AZ14170132.

DETAILED DESCRIPTION:
This is a non-randomized, open-label, fixed sequence study to be conducted at multiple study centers.

The study will consist of 2 parts:

Part A of the study will comprise of:

* Screening period
* Treatment period: The treatment period will comprise of Cycles 1, 2 and 3 where the participants will receive AZD5335 along with itraconazole
* Follow-up visit (not applicable for participants involved in Part B)

Part B of the study will comprise of:

* Treatment period: Cycle 4 and onwards
* Safety Follow-up period

ELIGIBILITY:
Inclusion Criteria:

* Participants with Platinum-resistant, relapsed, high- grade epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer and: (a) have received at least 1 prior line of platinum-containing chemotherapy and have progressed on or within 6 months after the date of the last dose of platinum; (b) must have received prior bevacizumab and/or Poly (ADP-ribose) polymerase (PARP) inhibitors according to local guidelines, unless ineligible.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.

Exclusion Criteria:

* Spinal cord compression or a history of leptomeningeal carcinomatosis.
* Unresolved toxicities of Grade ≥ 2 (National Cancer Institute-Common Terminology Criteria for Adverse Events v5.0) from prior therapy.
* History of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required oral or IV steroids or supplemental oxygen, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Uncontrolled intercurrent illness within 12 months prior to screening.
* Any other contraindication for receiving itraconazole according to the prescribing information and the Investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2027-10-22 (Estimated); Study Completion 2027-10-22 (Estimated)

PRIMARY OUTCOMES:
Area under curve from time 0 to time 17 days (AUC0-17days) | Cycle 2 and Cycle 3 (each cycle is of 21 days)
  The effect of itraconazole on the pharmacokinetics (PK) of AZ14170132 will be assessed.
Maximum plasma drug concentration (Cmax) | Cycle 2 and Cycle 3 (each cycle is of 21 days)
  The effect of itraconazole on the PK of AZ14170132 will be assessed.

SECONDARY OUTCOMES:
Maximum plasma drug concentration (Cmax) | Cycle 2 and Cycle 3 (each cycle is of 21 days)
  Cmax of AZ14170132 will be assessed.
Area under curve from time 0 to time 17 days (AUC0-17days) | Cycle 2 and Cycle 3 (each cycle is of 21 days)
  AUC0-17days of AZ14170132 will be assessed.
Minimum plasma drug concentration (Cmin) | Cycle 2 and Cycle 3 (each cycle is of 21 days)
  Cmin of AZ14170132 will be assessed.
Area under curve from time 0 to the time of last measurable concentration (AUC0-t) | Cycle 2 and Cycle 3 (each cycle is of 21 days)
  AUC0-t of AZ14170132 will be assessed.
Terminal elimination (lambda_z) | Cycle 2 and Cycle 3 (each cycle is of 21 days)
  lambda_z of AZ14170132 will be assessed.
Half life (t1/2) | Cycle 2 and Cycle 3 (each cycle is of 21 days)
  t1/2 of AZ14170132 will be assessed.
Time to maximum observed concentration (tmax) | Cycle 2 and Cycle 3 (each cycle is of 21 days)
  tmax of AZ14170132 will be assessed.
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Part A: up to 121 days; Part B: up to 365 days post last participant first dose
  The safety and tolerability of AZD5335 alone and in combination with itraconazole will be assessed.
Objective response rate (ORR) | Part A: up to 121 days; Part B: up to 365 days post last participant first dose
  The ORR is defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR), with the denominator defined as the number of participants in the response evaluable set.
Duration of response (DoR) | Part A: up to 121 days; Part B: up to 365 days post last participant first dose
  The DoR is defined as the time from the date of first documented objective response (which is subsequently confirmed) until date of first documented disease progression or death (by any cause in the absence of disease progression).
Progression-free Survival (PFS) | From Day 1 until until disease progression or death (up to 2 years)
  The PFS is defined as the time from the start of treatment until the date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the participant withdraws from randomised therapy or receives another anti-cancer therapy prior to progression.

CONTACTS AND LOCATIONS:
Locations (7):
- Georgia (2):
  - Research Site, Batumi
  - Research Site, Tbilisi
- Research Site, Dublin, Ireland
- Research Site, Lisbon, Portugal
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Logroño
  - Research Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure."Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitment a made to the EFPIA PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/